CLINICAL TRIAL: NCT00997997
Title: ARTOS - Avelox® in Routine Treatment of Complicated Skin and Skin Structure Infections
Brief Title: Avelox in Complicated Skin and Skin Structure Infections
Acronym: ARTOS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer HealthCare AG
Other Study IDs: 12237; 12236 (AX0502DE) (Other: Company); 12237 (AX0502AT) (Other: Company); 12519 (AX0502SI) (Other: Company); 12645 (AX0502BG) (Other: Company); 12646 (AX0502PK) (Other: Company); 12754 (AX0502GR) (Other: Company); 12865 (AX0502KR) (Other: Company); 12866 (AX0502TW) (Other: Company); 13045 (AX0502ID) (Other: Company); 13165 (AX0502PH) (Other: Company); 13206 (AX0502EG) (Other: Company); 13924 (AX0502SA) (Other: Company)
Record Dates: First submitted 2009-10-02; First posted 2009-10-20 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Skin Diseases, Bacterial
Keywords: Skin Diseases, Bacterial; Product Surveillance; Postmarketing
MeSH Terms: conditions — Skin Diseases, Bacterial | interventions — Moxifloxacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — 400 mg, intravenous / oral, once daily, treatment duration at the discretion of the attending physician who must consult the local product information

SUMMARY:
This international, prospective, non-interventional, non-controlled observational study obtains data on efficacy, safety and tolerability of Avelox treatment under daily-life treatment conditions. Specifically investigated are the improvement of clinical symptoms and the duration until infection improvement and cure.Any patient with a diagnosis of complicated skin and skin structure infection (cSSSI) treated with Avelox can be documented. The observation period for each subject covers the treatment period with Avelox. For each patient, the physician documents data at an initial visit and one or two follow-up visit(s) in line with routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a diagnosis of complicated skin and skin structure infection (cSSSI) and for whom the decision was made by the attending physician to start treatment with Avelox before inclusion into and independent of the study.

Exclusion Criteria:

* Exclusion criteria are those specified in the local product information.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients being diagnosed with complicated skin and skin structure infections, mainly in hospital settings
Sampling Method: Non-Probability Sample
Enrollment: 6127 (Actual)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Efficacy: course of severity of infection, course of clinical signs and symptoms, duration until improvement, duration until recovery, duration until wound closure, overall assessment of efficacy by the physician, reuse of Avelox | last documented follow-up visit, according to the respective praxis routine

SECONDARY OUTCOMES:
Adverse events collection | during entire study course, according to the respective praxis routine
Overall assessment of tolerability by the physician | last documented follow-up visit, according to the respective praxis routine

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (12):
- Many Locations, Austria
- Many Locations, Bulgaria
- Many Locations, Egypt
- Many Locations, Germany
- Many Locations, Greece
- Many Locations, Indonesia
- Many Locations, Pakistan
- Many Locations, Philippines
- Many Locations, Saudi Arabia
- Many Locations, Slovenia
- Many Locations, South Korea
- Many Locations, Taiwan